CLINICAL TRIAL: NCT05236933
Title: Association Between Types of Pain and Motor Activities Physical Activity in Individuals With Spinal Cord Injury
Brief Title: Association Between Types of Pain and Motor Activities Physical Activity
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 27219
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injury; Chronic Pain
Keywords: physical activity; virtual reality; nociceptive pain; neuropathic pain
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain; Motor Activity; Nociceptive Pain; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropathic: Individuals who report pain that is categorized as neuropathic will be assigned to this group.
- Nociceptive: Individuals who report pain that is categorized as nociceptive will be assigned to this group.

SUMMARY:
This study will investigate the relationships between: (1) physical activity (PA) and types of chronic pain (nociceptive and neuropathic), and (2) virtual reality (VR) and types of chronic pain (nociceptive and neuropathic).

DETAILED DESCRIPTION:
Chronic pain can be differentiated by its underlying mechanisms. However, this important distinction is not applied to most non-pharmacological treatment approaches. Studies that have shown modulation of chronic pain with physical activity (PA) or virtual reality (VR) have not evaluated differential effects on nociceptive and neuropathic pain. Therefore, it is unknown if neuropathic pain and nociceptive pain respond differently to PA and VR, and if treatment could be optimized through targeted interventions or a combination of interventions. Understanding the relationships between different types of pain and motor activity will provide new insight to inform future recommendations to alter PA levels for pain modulation.

A prospective, cohort design will be employed for this study of individuals with SCI for a duration of one week in the community. This study will identify trends that are different between the responses of different types of pain and motor activities (i.e., PA and VR). The data obtained will also capture fluctuations in PA levels across participants and corresponding pain levels because PA levels will be collected through real-world data in the community.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinal cord injury (SCI) (at least six months post-SCI)
* Experienced chronic pain for a duration of at least 6 months
* Functionally able to self-propel a manual wheelchair
* Medically stable

Exclusion Criteria:

* History of motion sickness or epilepsy
* Condition in which PA is medically contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic SCI who live in the Greater Philadelphia region and have experienced chronic pain are eligible to participate in the study. Recruitment efforts will be targeted equally towards men and women of all races and ethnicities, however because SCI is more prevalent in men, we anticipate higher recruitment of men than women.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity over 1 week | Measured repeatedly at set intervals; at baseline, 15 minutes after baseline assessment, and once daily for 1 week
  Patient-reported rating of pain intensity collected using the International SCI Pain Basic Data Set Version 2.0 (Widerstrom-Noga et al., 2014). This measure provides information regarding the location and severity of pain on a 0-10 scale, where higher number indicates worse pain, and categorization of pain into neuropathic and nociceptive.

SECONDARY OUTCOMES:
Pain interference | Measured once at baseline
  Pain interference will be collected using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference - Short Form 8a V1.0 (Amtmann et al., 2010). Pain interference is a measure of consequences of pain, rather than intensity. It incorporates aspects of pain associated with quality of life and physical functioning. A 5-point Likert scale for eight items provides a score ranging from 8-40, where a higher score indicates greater pain interference.
Depression | Measured once at baseline
  Depression will be measured using the Patient Health Questionnaire to examine its effect as a potential confounder in the interaction between physical activity and pain. This measure implements a 4-point Likert scale for nine items to calculate a score ranging from 0-27, with 0 indicating no depression and 27 indicating severe depression.
Kinesiophobia | Measured once at baseline
  The Tampa Scale for Kinesiophobia will be used in assessing kinesiophobia, which will assist in identifying if it is a confounder. This 17-item measure uses a 4-point Likert scale to calculate a score between 17-68, where higher scores indicate greater fear of movement.
Conditioned pain modulation | Measured once at baseline
  Conditioned pain modulation (CPM) is used to assess endogenous pain inhibition mechanisms. The outcome of CPM testing is either a normal effect or an abnormal effect. Abnormal CPM effect, which is an increased pain threshold after a conditioning stimulus, is an important biomarker of chronic pain (Fernandes et al., 2019).
Virtual embodiment | Measured once at baseline
  The Virtual Embodiment Questionnaire (Roth & Latoschik, 2020) will be used to assess embodiment with the avatar while in the immersive VR environment. This measure uses a 7-point Likert scale to calculate a score ranging from 4-28 in each of three sections that assess body ownership of the avatar, control and agency of the avatar, and sensation of body changes with the avatar. A higher score in each section indicates increased ownership, increased control, and increased body change, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Canori A, Coffman DL, Wright WG, Finley MA, Hiremath SV. Differential relationships between physical activity and pain phenotypes in individuals with spinal cord injury. J Spinal Cord Med. 2025 Jul;48(4):720-729. doi: 10.1080/10790268.2024.2344315. Epub 2024 Apr 25. PMID 38661677